CLINICAL TRIAL: NCT01313260
Title: Structural and Functional Connectivity in Partial Epilepsies Studied with MRI and MEG
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C09-21; 2010-A00399-30 (Registry Identifier: IDRCB)
Record Dates: First submitted 2011-02-15; First posted 2011-03-11 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Epilepsies
Keywords: Refractory partial epilepsies
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Epilepsy patients: Epilepsy patients selected before undergoing intracranial EEG recordings
- control group: Healthy volunteers

SUMMARY:
Surgery may be an effective therapy for refractory focal epilepsies with a clear delineated focus but surgical benefits are less clear for patients with a poorly defined focus such as non lesional refractory partial epilepsies.

SEEG is considered the criterion standard to localize the epileptogenic zone (EZ) but the procedure is risky with a limited spatial sampling. The development of non-invasive neuroimaging alternatives is thus an important goal to improve EZ delineation and optimize SEEG procedures.

The main hypothesis of this research project is the existence of a network organization specific for each patient which allows the generation and propagation of epileptic activities. The investigators wish to explore this network using diffusion tensor MRI to study structural connectivity and MEG/FMRI to study functional connectivity. The investigators will apply tools from the theories of complex networks and dynamical systems to characterize the network organization of epileptic process.

The investigators aimed to identify and localize differences in connectivity parameters between individual patients and a control group of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* intracranial EEG recordings scheduled
* no neurological or psychiatric disease for healthy volunteers

Exclusion Criteria:

* contraindication to MRI
* pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Refractory partial epilepsy patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-04-05 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Epileptic network assessed using structural and functional connectivity measures obtained with MRI and MEG | one year
  Structural connectivity will be assessed using diffusion tensor MRI including the following parameters: mean diffusivity and anisotropy at voxel level, fiber tractography.
  Functional connectivity will be assessed using Rs-FMRI or MEG signal correlation measures. Cortical parcellation will allow the location of connectivity parameters calculated using the graph theory.
  Structural and functional data from one given patient will be statistically compared those of the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- ICM (Brain and Spine Institute), Paris, France

REFERENCES:
- [Background] Chavez M, Valencia M, Navarro V, Latora V, Martinerie J. Functional modularity of background activities in normal and epileptic brain networks. Phys Rev Lett. 2010 Mar 19;104(11):118701. doi: 10.1103/PhysRevLett.104.118701. Epub 2010 Mar 18. PMID 20366507
- See also: Organization — http://www.inserm.fr/